CLINICAL TRIAL: NCT00694070
Title: Evaluation of a Diabetes Data Management System In a Clinical Setting
Brief Title: Evaluation of a Diabetes Data Management System
Status: Completed | Type: Observational
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: CTD-2008-11
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Results first posted 2009-09-23 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- health care professionals and lay users: h= 8 health care professionals p= 43 lay users

SUMMARY:
The purpose of this study is to evaluate a diabetes data management program in the hands of potential users, both health care professionals and lay users.

DETAILED DESCRIPTION:
Diabetes data management programs analyze blood glucose results downloaded from glucose meters to assist health care professionals or lay users manage their diabetes. During the study, subjects download meters, generate and print reports, evaluate the program's ease of use, and verify that they understand the program output.

ELIGIBILITY:
Inclusion Criteria:

* Health Care Professionals:

  1. Must have experience using diabetes data management software in the medical office such as downloading meters, reviewing reports (computer screen or printouts), or assisting in patients' diabetes disease management using software.
  2. May include: endocrinologists, primary care physicians, nurse educators, or other medical staff involved in downloading meters or interpreting the data output.
* Lay users must:

  1. Be at least 18 years of age.
  2. Have diabetes (or be the parent or legal guardian of a child with diabetes) and have been testing blood sugar at home at least twice daily for one month or more.
  3. Be able to speak, read and understand English.
  4. Currently using diabetes management software at home or be familiar with diabetes management software. At least 75% of subjects must have been using software for at least one month.
  5. Have experience using PC programs or browsing the internet.

Exclusion Criteria:

* Persons working for a competitive medical device company.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lay users males or females and health care professionals.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2008-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute
Locations (1):
- AMCR Institute, Escondido, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Health Care Professionals and Lay Users
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Health Care Professionals and Lay Users
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 53 [18 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Rated 80% of Tasks as Very Simple, Simple, or Neither Simple Nor Difficult (Ease of Use of the Software Program)
Description: After completing each task, subjects rated the ease of performing each task on a scale of 1 to 5.
  1. Very Simple
  2. Simple
  3. Neither simple nor difficult
  4. Difficult
  5. Very Difficult Outcome measure was the number of participants that rated 80% of tasks as 1,2, or 3.
Time Frame: 1-2 hours
Population: per protocol
Measure: Number; unit: Participants
Arm/Group | Health Care Professionals and Lay Users
Number analyzed (Participants) | 51
Participants | 46
Statistical Analysis 1: Comparison: Health Care Professionals and Lay Users; Test type: Non-Inferiority or Equivalence — The null and alternative hypotheses for these tests will have the form: Ho: Pr{Success} < Po vs. Ha: Pr{Success} ≥ Po. Critical values for numbers of successes were computed to give approximately a 90% chance of rejecting Ho in favor of the alternative (non-inferiority) if the true probability of success is at least Po. For Po = 80%, with n=51, critical number is 38. With this critical value and sample size, the power to reject Ho is approximately 87.43%; p = 0.0421, Exact binomial test

2. Primary Outcome: Number of Participants Rated as <= 3 (Success in Using the Program)
Description: Subjects were rated by study staff as to their success at performing basic tasks. The rating scale was:
  1. successful
  2. successful after being referred to user instructions
  3. success with assistance (similar to a customer call)
  4. unsuccessful 5 = software problem Outcome measure was the number of participants rated as <= 3.
Time Frame: 1-2 hours
Measure: Number; unit: Participants
Arm/Group | Health Care Professionals and Lay Users
Number analyzed (Participants) | 51
Participants | 50
Statistical Analysis 1: Comparison: Health Care Professionals and Lay Users; Test type: Non-Inferiority or Equivalence — The null and alternative hypotheses for these tests will have the form: Ho: Pr{Success} < Po vs. Ha: Pr{Success} ≥ Po. Critical values for numbers of successes were computed to give approximately a 90% chance of rejecting Ho in favor of the alternative (non-inferiority) if the true probability of success is at least Po. For Po = 95%, with n=51, critical number is 47. With this critical value and sample size, the power to reject Ho is approximately 88.96%; p = 0.0309, Exact binomial test

3. Primary Outcome: Number of Participants That Could Answer at Least 85% of the Comprehension Questions Correctly (Comprehension of the Program Reports)
Description: Subjects were asked thirty questions throughout the evaluation to test whether they understood the data displays, graphs and features of the software. Outcome measure was the number of participants that could answer at least 85% of the comprehension questions correctly.
Time Frame: 1-2 hours
Measure: Number; unit: participants
Arm/Group | Health Care Professionals and Lay Users
Number analyzed (Participants) | 51
participants | 50
Statistical Analysis 1: Comparison: Health Care Professionals and Lay Users; Test type: Non-Inferiority or Equivalence — The null and alternative hypotheses for these tests will have the form: Ho: Pr{Success} < Po vs. Ha: Pr{Success} ≥ Po. Critical values for numbers of successes were computed to give approximately a 90% chance of rejecting Ho in favor of the alternative (non-inferiority) if the true probability of success is at least Po. For Po = 90%, with n=51, critical number is 43. With this critical value and sample size, the power to reject Ho is approximately 93.57%; p = 0.0309, Exact binomial test

ADVERSE EVENTS:
Arm/Group | Health Care Professionals and Lay Users
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No